CLINICAL TRIAL: NCT01603784
Title: Combining Exercise and Cognitive Training to Improve Everyday Function
Acronym: EXACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: St. Louis Jewish Community Center (Unknown); St. Louis Naturally Occurring Retirement Community (NORC) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 201102416; 1R01AG034581-01 (NIH)
Record Dates: First submitted 2012-05-02; First posted 2012-05-23 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Effect of Exercise on Cognitive Function
Keywords: exercise; cognition; memory; adult
MeSH Terms: conditions — Motor Activity | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Combined (Experimental): Aerobic Exercise + Cognitive Training
  Interventions: Behavioral: Intensive Exercise; Behavioral: Cognitive Training
- Exercise (Experimental): Aerobic Exercise + Health Education
  Interventions: Behavioral: Intensive Exercise; Behavioral: Health Education
- Cognitive (Experimental): Home Exercise + Cognitive Training
  Interventions: Behavioral: Home Exercise; Behavioral: Cognitive Training
- Control (Experimental): Home Exercise + Health Education
  Interventions: Behavioral: Home Exercise; Behavioral: Health Education

INTERVENTIONS:
Behavioral: Intensive Exercise — Standardized aerobic training program that is individualized to each participant's fitness level, and supervised by a certified exercise specialist. Participants attend 3 training sessions per week for 6 months. The session begins with a 10-15 minute warm-up. Participants then exercise on a treadmill or stationary bike, followed by "cool-down" activities. Heart rate and rating of perceived exertion are used to evaluate exercise intensity. Participants begin at ~30 min/day 60-70% of HR max and/or an equivalent level of RPE, and progress to 45-50 minutes at 75-85% for HR max.
  Arms: Combined; Exercise
Behavioral: Home Exercise — Exercise program consisting of stretching, range of motion, and simple yoga exercises designed to improve flexibility. Each participant has a 60-minute sessions with an exercise trainer to teach them how to perform the exercises correctly. They are also given diagrams illustrating the exercises, along with written instructions. They are instructed to perform these exercises at home at least 3 times per week for 30 - 45 minutes. They also go to the recreational center monthly to meet with an exercise trainer to ensure that they are doing the exercises correctly. Participants record their exercise activities on a calendar for the 6 months.
  Arms: Cognitive; Control
Behavioral: Cognitive Training — Computer-based training that is is administered 3 days per week for 8 weeks during months 5 and 6. The training program focuses on 3 types of cognitive processes: task coordination, prospective memory, and retrospective memory retrieval. One day of the week is devoted to each of the three cognitive processes. Some training sessions include a homework assignment for application and practice of the target cognitive processes in everyday activities.
  Arms: Cognitive; Combined
Behavioral: Health Education — Weekly educational sessions are administered during months 5 and 6, conducted at the recreational center by research staff. Sessions last 1 hour, and cover health and other topics unrelated to exercise or cognition, such as nutrition, hearing loss, stroke, and saving energy in one's home. At the completion of each session, participants are given a "homework" assignment.
  Arms: Control; Exercise

SUMMARY:
The purpose of this randomized, controlled, prospective study is to evaluate the benefits of combining aerobic exercise with cognitive training for optimizing cognitive function. The study will enroll 109 men and women, age 55-75 years who are in stable health and without contraindications to exercise or evidence of dementia or cognitive impairment. Individuals will be randomly assigned to one of four groups for six months: Aerobic Exercise and Health Education, Home Exercise and Cognitive Training, Aerobic Exercise and Cognitive Training, and Home Exercise and Health Education. Participants will undergo measurements of cognitive function, physical performance, and complete questionaires about daily activities, physical activity, and quality of life at baseline (pre-intervention), and at 6 and 12 months after baseline.

ELIGIBILITY:
Inclusion Criteria:

* age 55-75 years (inclusive)
* English-speaking
* sufficient visual and auditory perception to complete testing
* available informant (someone who knows the individual well)
* Clinical Dementia Rating of 0 (non-demented per the screening assessment).

Exclusion Criteria:

* participation in a regular exercise program in last 6 months
* participation in a cognitive training program in last 6 months
* inability to walk on a treadmill or ride an exercise bike
* less than a 10th grade education
* mild cognitive impairment or dementia
* cigarette smoking within the previous year
* history of alcohol or substance abuse
* BMI greater than 35
* insulin-dependent diabetes
* major and/or unstable medical, neurological, or psychiatric disorder, including:

  * active congestive heart failure
  * unstable angina
  * effort angina
  * nocturnal angina
  * MI within previous 6 months
  * ECG evidence of serious arrhythmias and/or acute myocardial ischemia reflected by ST-segment depression of 0.3 mm
  * resting blood pressure above 170 systolic or 100 diastolic
  * chronic infections
  * advanced arthritis
  * contractures or weakness due to CVA that would prevent adequate performance of the exercises.
  * disabling stroke
  * late stage renal or liver disease
  * major affective disorder with active symptoms

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2010-03; Primary Completion 2012-08 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Memory for Medical Information | Change in memory task performance between baseline and 6 months
  This task measures the ability of the individual to learn and recall complex medical information, and the source of the information.
Cooking Breakfast task | Change in task performance between baseline and 6 months
  Participants engage in a computerized laboratory simulation of a cooking task to assesses cognitive dimensions of planning, prospective memory, monitoring the progress of ongoing activity, anticipating potential problems, task switching, and task coordination.
Virtual Week task | Change in task performance between baseline and 6 months
  Participants engage a computerized board game that simulates choices about, and recall of, daily and weekly activities.

SECONDARY OUTCOMES:
Activities of Daily Living--Yale Physical Activity Scale (YPAS) | Baseline, Month 3, Month 6, Month 12
  Questionnaire that objectively measures frequency and time spent per week performing common physical activities, which are used to caculate total weekly metabolic work (KCals).
Uniform Data Set (UDS) | Baseline, Month 12
  A standardized interview to ascertain and assess demographic information, health status, cognitive status, medications, and functional status. The interview is conducted with the research participant and a collateral source historian.
Geriatric Depression Scale | Baseline, Month 12
  A 15-item questionnaire to assess for symptoms of depression.
Late Life Function & Disability Index (LLFDI) | Baseline, Month 6, Month 12
  A standardized questionnaire to assess performance of activities of daily living (ADLs) and the level of difficulty experienced while performing each activity.
Pittsburgh Sleep Quality Index (PSQI) | Baseline, Month 6, Month 12
  Questionnaire to assess sleep quality and events in the prior month. Includes a section for roommate/bed partner response.
Objective Physical Performance Tests | Baseline, Month 6
  Physical Performance Test, Senior Fit Test, Dual Task Walking Speed. These tests objectively measure walking speed, muscle strength, balance, and coordination.
Prospective and Retrospective Memory Questionnaire (PMRQ) | Baseline, Month 6, Month 12
  Objective questionnaires to measure ability to learn and recall information.
Peak Aerobic Power | Baseline, Month 6
  The participant walks on a treadmill, with a progressively increased grade (level of incline)over a 8-15 minute period, with continuous measurements of expired oxygen and carbon dioxide. Information obtained is used to measure the total amount of work that the person performs during the test. The participant has continuous ECG monitoring during the test.
Cognitive assessment battery | Baseline, Month 6, Month 12
  Array of cognitive tasks to assess performance in a variety of areas. Includes Stroop (response time and attentional control), Trials A/B (sequencing), Crossing Off (motor control), Logical Memory (story recall), and Digit Symbol (corresponding symbols to digits).

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Binder, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States